CLINICAL TRIAL: NCT00500903
Title: An Open-Label, Dose Escalation Phase 1 Study of MLN8237, a Novel Aurora A Kinase Inhibitor, in Patients With Advanced Solid Tumors
Brief Title: A Study of MLN8237, a Novel Aurora A Kinase Inhibitor, in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C14001; U1111-1187-1087 (Registry Identifier: WHO)
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Advanced Malignancies
Keywords: Drug therapy
MeSH Terms: interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PIC Dose Escalation (Experimental): Alisertib 5, 10, 20, 40, 80, 110 or 150 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 7 to 21 days followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib--related toxicity (up to 51 cycles).
  Interventions: Drug: Alisertib
- ECT Dose Escalation (Experimental): Alisertib 10 or 20 mg, Enteric-coated Tablet (ECT) formulation, orally, once daily (QD) for 7 days followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib--related toxicity (up to 2 cycles).
  Interventions: Drug: Alisertib
- Relative Bioavailability (Experimental): Alisertib 40 mg ECT or PIC formulation, orally, twice daily (BID) for 7 days followed by a 14--day recovery period in cycle 1, followed by alisertib 40 mg in the opposite formulation (PIC or ECT) orally, twice daily (BID) for 7 days followed by a 14--day recovery period in cycle 2, followed by alisertib 50 mg PIC formulation orally, twice daily (BID) for 7 days followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib--related toxicity (up to 9 cycles).
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib (MLN8237) will be supplied in capsules of 5 or 25 mg and will be given on an empty stomach, with patients remaining nothing by mouth except for water and prescribed medications for 2 hours before and 1 hour after each dose. Each dose will be given by mouth with 8 ounces of water for 7 to 21 consecutive days. A 14-day recovery period will follow each dosing period regardless of its duration.
  Other Names: MLN8237

SUMMARY:
To determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of MLN8237 when given by mouth (PO) for a minimum of 7 and a maximum of 21 consecutive days, followed by a 14-day recovery period.

DETAILED DESCRIPTION:
The drug tested in this study is called alisertib. Alisertib is being tested to treat people who have advanced malignancies. This study determined the dose-limiting toxicity, maximum tolerated dose, safety and pharmacokinetics (how the drug moves through the body) for alisertib when given once or twice a day for 7 to 21 days. This open label study enrolled 87 participants. Participants were enrolled in one of 3 treatment groups:

* Powder-in-Capsule (PIC) Dose Escalation (alisertib 5, 10, 20, 40, 80, 110 or 150 mg PIC , once daily (QD) for 7 days (D),or alisertib 25 mg, PIC, orally, QD 14D, or alisertib 25, 50 or 70 mg, PIC, orally, QD 21D, or alisertib 50 or 60 mg, PIC, orally, twice daily (BID) 7D, alisertib 40 mg, PIC, orally, BID 14D
* ECT Dose Escalation (alisertib 10 or 20 mg, Enteric-coated Tablets (ECT), orally, QD for 7 to 21 days
* Relative Bioavailability (alisertib 40 mg ECT or PIC, orally, BID 7D in cycle 1, followed by alisertib 40 mg in the opposite formulation (PIC or ECT) orally, BID 7D in cycle 2, followed by alisertib 50 mg PIC orally, BID 7D in each additional All participants received treatment until their disease progressed or they experienced unacceptable alisertib-related toxicity. This multi-center trial was conducted in the United States. The overall time to participate in this study was 1011 days. Participants made multiple visits to the clinic, including a final visit 30 days after receiving their last dose of alisertib for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic and/or advanced solid tumors (including lymphomas) for which no effective standard treatment is available
* Aged 18 years or more
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Expected survival longer than 3 months from enrollment in the study
* Radiographically or clinically evaluable tumor; however, measurable disease as defined by (RECIST) criteria is not required for participation in this study
* Suitable venous access for the conduct of blood sampling for MLN8237 PK
* Recovered from the reversible effects of prior antineoplastic therapy (with the exception of alopecia and grade 1 neuropathy) with at least 4 weeks elapsed since the last exposure to cytotoxic chemotherapy or to radiotherapy and at least 6 weeks elapsed since exposure to nitrosoureas or mitomycin C. Participants treated with fully human monoclonal antibodies must not have received treatment with such antibodies for at least 6 weeks, and those treated with chimeric monoclonal antibodies must not have received treatment with such antibodies for at least 4 weeks. Participants treated with noncytotoxic small molecule drugs (eg, tyrosine kinase inhibitors, such as Tarceva®, and hormonal agents, such as Femara®) must not have received treatment with these drugs for at least 2 weeks before the first dose of MLN8237 is given.
* Male participants must use an appropriate method of barrier contraception (eg, condoms) and inform any sexual partners that they must also use a reliable method of contraception (eg, birth control pills) from the time of informed consent until 3 months after the last dose of study treatment.
* Female participants must be postmenopausal, surgically sterilized, or willing to use reliable methods of birth control (eg, a hormonal contraceptive, an intrauterine device, diaphragm with spermicide, or abstinence) and inform male sexual partners that they must also use a reliable method of contraception (eg, condoms) from the time of informed consent until 3 months after the last dose of study treatment.
* Willing and able to give written informed consent before the conduct of any study related procedure that is not part of normal medical care, and willing to comply with the protocol

Exclusion Criteria:

* Pregnant or lactating
* Major surgery or serious infection within the 28 days preceding the first dose of study treatment
* Life-threatening illness or uncontrolled medical illness unrelated to cancer
* Ongoing nausea or vomiting of any severity
* > Grade 1 diarrhea
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of MLN8237. Examples include but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease.
* History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease.
* Difficulty swallowing capsules
* Inability to take nothing by mouth except for water and prescribed medications for 2 hours before and 1 hour after each dose of MLN8237
* Received more than 4 previous cytotoxic chemotherapeutic regimens including regimens used as adjuvant or neo-adjuvant therapies. There is no limit on the number of noncytotoxic therapies (eg, hormonal and immunologic) that participants may have received. Tyrosine kinase inhibitors (eg, Tarceva and Iressa®) are considered noncytotoxic compounds.
* Prior treatment with high-dose chemotherapy, defined as chemotherapy requiring the use of peripheral blood or bone marrow stem cell support for hematopoietic reconstitution
* Prior treatment with radiation therapy involving ≥25% of the hematopoietically active bone marrow
* Clinical and/or radiographic evidence of cerebral metastases. However, participants who have a history of central nervous system (CNS) metastasis but who have no radiographic or clinical evidence of residual tumor (eg, following complete surgical resection or stereotactic radiosurgery) are not excluded from participation in this study
* Absolute neutrophil count <1500/mm^3; platelet count <100,000/mm^3
* Serum creatinine >1.6 mg/dl or a measured or estimated creatinine clearance <40 mL/minute
* Bilirubin >1.5 times the upper limit of the normal range (ULN); aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >2.5 times the ULN, and alkaline phosphatase (ALP) >2.5 times the ULN. Both the AST and ALP may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of metastatic disease to liver and/or to bone; however, the ALT must in all circumstances be <2.5 times the ULN
* Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinically significant or baseline prolongation of the rate-corrected QT interval (eg, repeated demonstration of QTc interval > 450 milliseconds)
* Left ventricular ejection fraction (LVEF) < 50%
* Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection. Testing for these agents is not required in the absence of clinical findings or suspicion.
* Less than 4 weeks between the last dose of an investigational agent and the first dose of MLN8237
* Admission or evidence of benzodiazepine dependence or abuse and/or alcohol abuse or an inability to restrict consumption of alcohol to no more than 1 standard unit of alcohol per day during the study and for 30 days from the last dose of study treatment. A standard unit of alcohol is defined as one 12-oz (150mL) beer, 1.5 oz (45mL) of 80-proof alcohol, or one 6-oz (175mL) glass of wine.
* Lactose intolerant, for the food effect cohort only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-05-15 (Actual); Primary Completion 2010-08-01 (Actual); Study Completion 2011-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Sarah Cannon Research Institute (SCRI), Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 15 May 2007 to 23 February 2011.
Pre-assignment Details: Participants with a diagnosis of advanced malignancies were enrolled in 1 of 3 treatment groups, alisertib 5 to 150 mg Powder-in-Capsule (PIC) dose escalation cohort, alisertib 10 or 20 mg Enteric-coated Tablet (ECT) dose escalation cohort, or alisertib 40 mg PIC/ECT in a crossover design followed by alisertib 50 mg relative bioavailability cohort.
Groups:
- PIC Dose Escalation: Alisertib 5, 10, 20, 40, 80, 110 or 150 mg, PIC, orally, once daily (QD) for 7 days, followed by a 14-day recovery period or alisertib 25 mg, PIC, orally, QD for 14 days, followed by a 14-day recovery period or alisertib 25, 50 or 70 mg, PIC, orally, QD for 21 days followed by a 14-day recovery period or alisertib 50 or 60 mg, PIC, orally, twice daily (BID) for 7 days followed by a 14-day recovery period or alisertib 40 mg, PIC, orally, BID for 14 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 51 cycles).
Period: Overall Study
Arm/Group | PIC Dose Escalation | ECT Dose Escalation | Relative Bioavailability
Started | 65 | 2 | 20
Completed | 0 | 0 | 0
Not Completed | 65 | 2 | 20
Not completed — Occurrence of Adverse Event(s) | 10 | 0 | 0
Not completed — Unsatisfactory Therapeutic Response | 2 | 0 | 0
Not completed — Progressive Disease | 41 | 2 | 15
Not completed — Patient Declined Further Treatment | 0 | 0 | 3
Not completed — Symptomatic Deterioration | 2 | 0 | 0
Not completed — Reason Not Specified | 10 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PIC Dose Escalation | ECT Dose Escalation | Relative Bioavailability | Total
Number analyzed (Participants) | 65 | 2 | 20 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.44) | 57.0 (15.56) | 56.9 (11.71) | 60.4 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 1 | 9 | 43
  Male | 32 | 1 | 11 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 56 | 2 | 20 | 78
  Not Reported | 7 | 0 | 0 | 7
  Hispanic or Latino | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 55 | 2 | 18 | 75
  Black or African American | 9 | 0 | 2 | 11
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 65 | 2 | 20 | 87
Height [Mean (Standard Deviation); unit: cm] | 169.3 (10.06) | 165.1 (0.00) | 171.5 (12.51) | 169.7 (10.55)
Weight [Mean (Standard Deviation); unit: kg] | 78.24 (18.130) | 67.36 (11.226) | 83.97 (21.706) | 79.33 (18.976)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — BSA=square root[height (cm) x weight (kg)/3600]
  m^2 | 1.91 (0.263) | 1.75 (0.147) | 1.99 (0.294) | 1.92 (0.270)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT was evaluated according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 and was defined as any of the following events related to therapy with alisertib:
  1. Grade 4 neutropenia lasting ≥7 consecutive days
  2. Grade 4 neutropenia with fever and/or infection
  3. Platelet count <25,000/mm^3
  4. Grade 3 or greater nausea and/or emesis despite use of optimal antiemetic prophylaxis
  5. Grade 3 or greater diarrhea despite maximal supportive therapy with loperamide
  6. Any other Grade 3 or greater nonhematologic toxicity, with the following exceptions: Grade 3 arthralgia/myalgias, Any grade of alopecia, Brief (<1 week) Grade 3 fatigue
  7. Treatment delay of >1 week due to failure of adequate hematologic or nonhematologic recovery from previous cycle of treatment
  8. Other alisertib-related nonhematologic toxicities ≥Grade 2 that, in the opinion of the investigator, required a dose reduction or discontinuation of therapy with alisertib.
Time Frame: Cycle 1 Day 1 up to Day 35 (alisertib daily for 7 to 21 days followed by a 14-day recovery period)
Population: DLT-Evaluable Population included all participants who received at least 75% of their planned alisertib doses for their first cycle of treatment (unless interrupted by DLT) and had sufficient follow-up data to allow the investigators and sponsor to determine whether DLT occurred.
Measure: Number; unit: participants
Groups:
- Alisertib 5 mg PIC QD 7D: Alisertib 5 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 4 cycles).
- Alisertib 10 mg PIC QD 7D: Alisertib 10 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 5 cycles).
- Alisertib 20 mg PIC QD 7D: Alisertib 20 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 31 cycles).
- Alisertib 40 mg PIC QD 7D: Alisertib 40 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 8 cycles).
- Alisertib 80 mg PIC QD 7D: Alisertib 80 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 15 cycles).
- Alisertib 110 mg PIC QD 7D: Alisertib 110 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles).
- Alisertib 150 mg PIC QD 7D: Alisertib 150 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 51 cycles).
- Alisertib 25 mg PIC QD 14D: Alisertib 25 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 14 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 5 cycles).
- Alisertib 25 mg PIC QD 21D: Alisertib 25 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 21 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles).
- Alisertib 50 mg PIC QD 21D: Alisertib 50 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 21 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 7 cycles).
- Alisertib 70 mg PIC QD 21D: Alisertib 70 mg, Powder-in-Capsule (PIC), orally, once daily (QD) for 21 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles).
- Alisertib 50 mg PIC BID 7D: Alisertib 50 mg, Powder-in-Capsule (PIC), orally, twice daily (BID) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 4 cycles).
- Alisertib 60 mg PIC BID 7D: Alisertib 60 mg, Powder-in-Capsule (PIC), orally, twice daily (BID) for 7 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 35 cycles).
- Alisertib 40 mg PIC BID 14D: Alisertib 40 mg, Powder-in-Capsule (PIC), orally, twice daily (BID) for 14 days (D) followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles).
- Alisertib 10 mg ECT QD7: Alisertib 10 mg, Enteric-coated Tablet (ECT) formulation, orally, once daily (QD) for 7 days followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib--related toxicity (up to 2 cycles).
- Alisertib 20 mg ECT QD7: Alisertib 20 mg, Enteric-coated Tablet (ECT) formulation, orally, once daily (QD) for 7 days followed by a 14--day recovery period in each cycle until disease progression or unacceptable alisertib--related toxicity (up to 2 cycles).
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D | Alisertib 25 mg PIC QD 14D | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D | Alisertib 40 mg PIC BID 14D | Alisertib 10 mg ECT QD7 | Alisertib 20 mg ECT QD7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 7 | 11 | 6 | 2 | 1 | 1
participants | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Alisertib
Description: MTD was defined as the highest dose at which DLT occurred in 0/3 or 1/6 patients.
Time Frame: From first dose of study drug to 30 days after the last dose (up to 1011 days)
Population: as for outcome 1
Measure: Number; unit: mg BID for 7 Days
Groups:
- Alisertib: Alisertib 5, 10, 20, 40, 80, 110 or 150 mg, PIC, orally, once daily (QD) for 7 days, followed by a 14-day recovery period or alisertib 25 mg, PIC, orally, QD for 14 days, followed by a 14-day recovery period or alisertib 25, 50 or 70 mg, PIC, orally, QD for 21 days followed by a 14-day recovery period or alisertib 50 or 60 mg, PIC, orally, twice daily (BID) for 7 days followed by a 14-day recovery period or alisertib 40 mg, PIC, orally, BID for 14 days followed by a 14-day recovery period or alisertib 10 or 20 mg ECT, orally QD for 7 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 51 cycles).
Arm/Group | Alisertib
Number analyzed (Participants) | 65
mg BID for 7 Days | 50

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From first dose of study drug to 30 days after the last dose (up to 1011 days)
Population: Safety Population included all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | PIC Dose Escalation | ECT Dose Escalation | Relative Bioavailability
Number analyzed (Participants) | 65 | 2 | 20
participants
  AEs | 65 | 2 | 20
  SAEs | 26 | 0 | 1

4. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose and Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: Pharmacokinetic (PK)-Evaluable Population included all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6
nM
  Day 1 | 208.4 (27.96) | 279.1 (46.20) | 759.3 (11.82) | 1245.4 (20.60) | 1661.3 (45.20) | 2717.8 (44.62) | 4260.3 (42.62)
  Day 7: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 6 | 5
  Day 7 | 285.7 (32.74) | 931.5 (81.68) | 1114.1 (36.96) | 1681.6 (64.62) | 2376.3 (51.06) | 3586.4 (48.28) | 4467.8 (24.58)

5. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6
hours (h)
  Day 1 | 2.000 [1.50 to 3.00] | 2.000 [1.50 to 3.00] | 1.500 [1.50 to 1.50] | 2.000 [1.50 to 6.00] | 2.000 [1.50 to 3.00] | 2.000 [1.48 to 5.57] | 2.000 [1.45 to 3.00]
  Day 7: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 6 | 5
  Day 7 | 1.500 [1.00 to 1.50] | 3.750 [1.50 to 6.00] | 1.500 [1.50 to 2.00] | 2.000 [1.97 to 6.00] | 2.000 [1.98 to 3.05] | 3.710 [1.42 to 6.02] | 2.000 [1.48 to 3.93]

6. Secondary Outcome: AUCt: Area Under the Concentration-Time Curve From Time 0 to Time t for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6
nM*h
  Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 6 | 6
  Day 1 | 1682.4 (31.06) | 2525.8 (21.87) | 5772.1 (10.68) | 12045.4 (57.01) | 20958.1 (38.92) | 29460.7 (39.43) | 38582.1 (45.95)
  Day 7: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 6 | 5
  Day 7 | 2919.5 (32.31) | 10602.9 (107.87) | 10927.5 (45.27) | 21976.0 (96.64) | 27825.5 (53.59) | 46271.1 (33.38) | 53031.9 (26.22)

7. Secondary Outcome: Terminal Half-Life (t1/2) for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: Pharmacokinetic (PK)-Evaluable Population included all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 2 | 2 | 3 | 2 | 3 | 6 | 5
h | 24.950 (20.4354) | 35.150 (23.4052) | 26.400 (19.7684) | 18.155 (12.5087) | 39.333 (18.8006) | 13.427 (4.3465) | 16.766 (9.7804)

8. Secondary Outcome: Accumulation Ratio (Rac) for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 6 | 5
ratio | 1.753 (0.2754) | 6.350 (7.2408) | 2.037 (0.9708) | 1.997 (0.9393) | 1.535 (0.3323) | 1.677 (0.6788) | 1.588 (0.4129)

9. Secondary Outcome: Peak/Trough Ratio for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 6 | 5
ratio | 4.107 (0.8460) | 5.195 (3.9527) | 5.430 (2.4856) | 3.907 (2.3944) | 3.850 (2.0612) | 4.922 (2.5890) | 4.610 (0.5314)

10. Secondary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)/h
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 6 | 5
liters (L)/h | 3.302 (35.8915) | 1.817 (107.8347) | 3.525 (49.1267) | 3.511 (72.1346) | 5.545 (41.0258) | 4.348 (61.5266) | 5.450 (37.3021)

11. Secondary Outcome: Ae: Amount of Alisertib Excreted in Urine Over the Collection Period for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose
Population: Pharmacokinetic (PK)-Evaluable Population included all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis.
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 6 | 6
ng | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 4806.7 (8325.39) | 18815.0 (1675.84) | 13813.3 (16387.22) | 14473.3 (15603.71)

12. Secondary Outcome: CLr: Renal Clearance of Alisertib as Powder-in-Capsule (PIC) With Once Daily for 7 Days (QD7D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 1 | 1 | 5 | 5
L/h | 0.0012630 (NA) — Cannot be calculated for 1 participant | 0.0013860 (NA) — Cannot be calculated for 1 participant | 0.0009414 (0.00063956) | 0.0006710 (0.00060091)

13. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
nM
  Day 1 | 778.7 (24.28)
  Day 7 | 995.5 (43.21)
  Day 14 | 808.9 (37.96)

14. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
h
  Day 1 | 4.000 [2.00 to 8.88]
  Day 7 | 2.000 [2.00 to 2.00]
  Day 14 | 2.000 [1.098 to 2.00]

15. Secondary Outcome: AUCt: Area Under the Concentration--Time Curve From Time 0 to Time t for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
nM*h
  Day 1 | 8061.6 (17.30)
  Day 7 | 8634.0 (42.70)
  Day 14 | 8978.0 (20.15)

16. Secondary Outcome: Terminal Half-Life for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: Cycle 1 Day 14 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
h | 65.67 (43.859)

17. Secondary Outcome: Accumulation Ratio (Rac) for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: Cycle 1 Days 7 and 14 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
ratio
  Day 7 | 1.203 (0.6964)
  Day 14 | 1.133 (0.2303)

18. Secondary Outcome: Peak/Trough Ratio for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: Cycle 1 Days 7 and 14 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
ratio
  Day 7 | 6.877 (1.1151)
  Day 14 | 5.073 (2.2113)

19. Secondary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: Cycle 1 Days 7 and 14 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
L/h
  Day 7 | 6.030 (2.9963)
  Day 14 | 5.433 (0.9808)

20. Secondary Outcome: Ae: Amount of Alisertib Excreted in Urine Over the Collection Period for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
ng | 800.0 (1385.64)

21. Secondary Outcome: CLr: Renal Clearance of Alisertib as Powder-in-Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 1
L/h | 0.0004930 (NA) — Cannot be calculated for 1 participant

22. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints up to 24 hours postdose and Days 14 and 21 predose and at multiple time points (up to 10 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
nM
  Day 1 | 898.2 (86.35) | 1725.9 (54.70) | 2237.0 (54.18)
  Day 14: number analyzed (Participants) | 3 | 6 | 5
  Day 14 | 1343.3 (60.32) | 1722.0 (38.82) | 2598.3 (12.49)
  Day 21: number analyzed (Participants) | 3 | 6 | 5
  Day 21 | 1104.7 (45.15) | 1564.2 (38.80) | 1974.5 (59.49)

23. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: as for outcome 22
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
h
  Day 1 | 2.020 [2.00 to 4.00] | 2.285 [2.00 to 4.00] | 2.000 [2.00 to 2.02]
  Day 14: number analyzed (Participants) | 3 | 6 | 5
  Day 14 | 2.000 [2.00 to 2.18] | 2.000 [1.98 to 2.03] | 2.000 [2.00 to 2.05]
  Day 21: number analyzed (Participants) | 3 | 6 | 5
  Day 21 | 2.000 [1.00 to 2.02] | 2.000 [1.93 to 9.92] | 2.000 [1.00 to 6.00]

24. Secondary Outcome: AUCt: Area Under the Concentration-time Curve From Time 0 to Time t for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: as for outcome 22
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
nM*h
  Day 1: number analyzed (Participants) | 3 | 6 | 6
  Day 1 | 10058.0 (66.85) | 14686.6 (44.04) | 22114.8 (68.66)
  Day 14: number analyzed (Participants) | 3 | 6 | 4
  Day 14 | 15131.7 (49.89) | 17168.2 (32.09) | 23197.2 (17.75)
  Day 21: number analyzed (Participants) | 3 | 6 | 5
  Day 21 | 13199.3 (70.05) | 19336.3 (26.85) | 23499.8 (65.64)

25. Secondary Outcome: Terminal Half-Life (t1/2) for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: Cycle 1 Day 21 predose and at multiple time points (up to 10 hours) postdose
Population: Pharmacokinetic (PK)-Evaluable Population included all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 5
h | 31.667 (6.7122) | 23.650 (16.9487) | 22.378 (19.8802)

26. Secondary Outcome: Accumulation Ratio (Rac) for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: Cycle 1 Days 14 and 21 predose and at multiple timepoints (up to 10 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
ratio
  Day 14: number analyzed (Participants) | 3 | 6 | 3
  Day 14 | 1.560 (0.5543) | 1.230 (0.4193) | 1.440 (0.1493)
  Day 21: number analyzed (Participants) | 3 | 6 | 4
  Day 21 | 1.560 (1.0516) | 1.373 (0.4474) | 1.335 (0.4749)

27. Secondary Outcome: Peak/Trough Ratio for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: Cycle 1 Days 14 and 21 predose and at multiple timepoints up to 10 hours postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
ratio
  Day 14: number analyzed (Participants) | 3 | 6 | 5
  Day 14 | 4.773 (0.9001) | 7.543 (5.4982) | 6.392 (2.0824)
  Day 21: number analyzed (Participants) | 3 | 6 | 5
  Day 21 | 3.637 (1.8675) | 4.157 (2.1051) | 5.570 (2.5772)

28. Secondary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: Cycle 1 Days 14 and 21 predose and at multiple timepoints up to 10 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
L/h
  Day 14: number analyzed (Participants) | 3 | 6 | 4
  Day 14 | 3.181 (42.5706) | 5.612 (28.6881) | 5.825 (17.7291)
  Day 21: number analyzed (Participants) | 3 | 6 | 5
  Day 21 | 3.656 (89.5750) | 4.984 (25.6945) | 5.745 (42.3818)

29. Secondary Outcome: Ae: Amount of Alisertib Excreted in Urine Over the Collection Period for Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
ng | 3047.7 (5278.71) | 5766.7 (7971.95) | 9391.4 (11410.18)

30. Secondary Outcome: CLr: Renal Clearance of Alisertib as Powder-in-Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 1 | 3 | 4
L/h | 0.0008640 (NA) — Cannot be calculated for 1 participant | 0.0012323 (0.00111840) | 0.0007865 (0.00042447)

31. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 11 | 6
nM
  Day 1 | 1581.1 (37.34) | 1867.1 (29.03)
  Day 7: number analyzed (Participants) | 10 | 5
  Day 7 | 3376.4 (41.74) | 3080.8 (38.79)

32. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 11 | 6
h
  Day 1 | 2.000 [1.98 to 8.00] | 2.000 [1.60 to 4.00]
  Day 7: number analyzed (Participants) | 10 | 5
  Day 7 | 2.015 [0.98 to 6.05] | 2.000 [1.98 to 6.03]

33. Secondary Outcome: AUCt: Area Under the Concentration-time Curve From Time 0 to Time t for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 11 | 6
nM*h
  Day 1: number analyzed (Participants) | 8 | 3
  Day 1 | 11166.3 (37.45) | 13200.4 (26.70)
  Day 7: number analyzed (Participants) | 5 | 4
  Day 7 | 32291.5 (40.82) | 27386.1 (37.43)

34. Secondary Outcome: Terminal Half-Life (t1/2) for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: Cycle 1 Day 8
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 10 | 6
h | 20.215 (15.5083) | 18.200 (3.2212)

35. Secondary Outcome: Accumulation Ratio (Rac) for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 5 | 3
ratio | 2.474 (1.0467) | 2.543 (0.1950)

36. Secondary Outcome: Peak/Trough Ratio for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 6 | 4
ratio | 2.193 (1.1346) | 1.890 (0.2012)

37. Secondary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 5 | 4
L/h | 2.984 (43.8719) | 4.220 (47.9681)

38. Secondary Outcome: Ae: Amount of Alisertib Excreted in Urine Over the Collection Period for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 10 | 5
ng | 13775.0 (7937.14) | 8498.3 (6866.09)

39. Secondary Outcome: CLr: Renal Clearance of Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 7 Days (BID7D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 10 | 5
ng | 0.001 (0.0011) | 0.001 (0.0004)

40. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 14 Days (BID14D) Dosing
Time Frame: Cycle 1 Days 1 and 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 40 mg PIC BID 14D
Number analyzed (Participants) | 2
nM
  Day 1 | 1236.6 (37.29)
  Day 7: number analyzed (Participants) | 1
  Day 7 | 2060.0 (NA) — Geometric Coefficient of Variation cannot be calculated for 1 participant.

41. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 14 Days (BID14D) Dosing
Time Frame: Cycle 1 Days 1 and 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 40 mg PIC BID 14D
Number analyzed (Participants) | 2
h
  Day 1 | 3.00 [2.0 to 4.0]
  Day 7: number analyzed (Participants) | 1
  Day 7 | 1.70 [1.7 to 1.7]

42. Secondary Outcome: AUCt: Area Under the Concentration-time Curve From Time 0 to Time t for Alisertib as Powder-in-Capsule (PIC) With Twice Daily for 14 Days (BID14D) Dosing
Time Frame: Cycle 1 Day 1 predose and at multiple time-points (up to 24 hours) postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 40 mg PIC BID 14D
Number analyzed (Participants) | 2
nM*h | 9684.8 (71.50)

43. Secondary Outcome: AUCt: Area Under the Concentration-time Curve From Time 0 to Time t as Assessment of Relative Bioavailability for Alisertib as Enteric-coated Tablet (ECT) Versus PIC at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nM*h
Groups:
- Alisertib 40 mg ECT BID 7D: Alisertib 40 mg, Enteric-coated tablet (ECT), orally, twice daily (BID) for 7 days (D) followed by a 14--day recovery period for 1 cycle.
- Alisertib 40 mg PIC BID 7D: Alisertib 40 mg, Powder-in-Capsule (PIC), orally, twice daily (BID) for 7 days (D) followed by a 14--day recovery period for 1 cycle.
Arm/Group | Alisertib 40 mg ECT BID 7D | Alisertib 40 mg PIC BID 7D
Number analyzed (Participants) | 14 | 14
nM*h | 12700.0 (6557.58) | 14190.7 (7097.72)

44. Secondary Outcome: Cmax: Maximum Observed Concentration as Assessment of Relative Bioavailability for Alisertib as Enteric-coated Tablet (ECT) Versus PIC at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple time-points (up to 10 hours) postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Alisertib 40 mg ECT BID 7D | Alisertib 40 mg PIC BID 7D
Number analyzed (Participants) | 14 | 14
nM | 1666.1 (765.28) | 2027.9 (928.96)

45. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Mitotic Index With PIC Once Daily for 7 Days (QD7D) Dosing
Description: Mitotic index was defined as the mean number of mitotic cells per millimeter (mm) length of the basoepithelial layer (BEL). Mitotic cells were counted manually within the BEL of 4, 5 µM skin sections by staining with fluorescent-tagged antibodies specific to 2 mitotic markers-serine 10 phosphohistone H3 (pHistH3) and MPM2. Deoxyribonucleic acid (DNA) was stained with a fluorescent marker as well. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose
Population: Pharmacokinetic (PK)-Evaluable Population included all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available at the given time-points.
Measure: Mean (Standard Deviation); unit: mitotic cells/millimeter of BEL
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 5 | 6
mitotic cells/millimeter of BEL
  Day 1, Hour 6 | 0.405 (0.2701) | 0.614 (0.5437) | 0.263 (0.1461) | 0.168 (0.5146) | 0.488 (1.0215) | 0.261 (0.4597) | 0.865 (0.9420)
  Day 1, Hour 24 | 0.019 (0.1914) | -0.103 (0.0186) | 0.005 (0.0709) | 0.141 (0.3852) | 0.108 (0.4081) | 1.764 (2.6380) | 0.239 (0.6992)

46. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Apoptotic Index With PIC Once Daily for 7 Days (QD7D) Dosing
Description: Apoptotic index was defined as the mean number of apoptotic cells per millimeter (mm) length of the basoepithelial layer (BEL). Apoptotic cells were counted manually within the BEL of 4, 5 µM skin sections by staining with hematoxylin-eosin. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: apoptotic cells/millimeter of BEL
Arm/Group | Alisertib 5 mg PIC QD 7D | Alisertib 10 mg PIC QD 7D | Alisertib 20 mg PIC QD 7D | Alisertib 40 mg PIC QD 7D | Alisertib 80 mg PIC QD 7D | Alisertib 110 mg PIC QD 7D | Alisertib 150 mg PIC QD 7D
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 5 | 6
apoptotic cells/millimeter of BEL
  Day 1, Hour 6 | 0.010 (0.1175) | -0.090 (0.1278) | 0.042 (0.0731) | 0.040 (0.0701) | 0.121 (0.1317) | 0.036 (0.0530) | -0.042 (0.1262)
  Day 1, Hour 24 | 0.009 (0.1164) | 0.065 (0.1404) | 0.000 (0.0000) | 0.037 (0.0634) | 0.074 (0.1286) | 0.151 (0.1721) | 0.139 (0.2069)

47. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Mitotic Index With PIC Once Daily for 14 Days (QD14D) Dosing
Description: as for outcome 45
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: mitotic cells/millimeter of BEL
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
mitotic cells/millimeter of BEL
  Day 1, Hour 6 | 0.134 (0.1723)
  Day 1, Hour 24 | 0.047 (0.0589)

48. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Apoptotic Index With PIC Once Daily for 14 Days (QD14D) Dosing
Description: as for outcome 46
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: apoptotic cells/millimeter of BEL
Arm/Group | Alisertib 25 mg PIC QD 14D
Number analyzed (Participants) | 3
apoptotic cells/millimeter of BEL
  Day 1, Hour 6 | 0.000 (0.0000)
  Day 1, Hour 24 | 0.000 (0.0000)

49. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Mitotic Index With PIC Once Daily for 21 Days (QD21D) Dosing
Description: as for outcome 45
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose and Days 7 and 21, 6 hours postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mitotic cells/millimeter of BEL
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
mitotic cells/millimeter of BEL
  Day 1, Hour 6: number analyzed (Participants) | 3 | 3 | 1
  Day 1, Hour 6 | 0.380 (0.4165) | 0.405 (0.4690) | 0.510 (NA) — Cannot be calculated for 1 participant
  Day 1, Hour 24: number analyzed (Participants) | 3 | 3 | 2
  Day 1, Hour 24 | 0.021 (0.1081) | 0.082 (0.1796) | 0.289 (0.5746)
  Day 7, Hour 6: number analyzed (Participants) | 0 | 0 | 3
  Day 7, Hour 6 |  |  | 0.479 (0.3040)
  Day 21, Hour 6: number analyzed (Participants) | 0 | 1 | 3
  Day 21, Hour 6 |  | 0.045 (NA) — Cannot be calculated for 1 participant. | 0.742 (0.5782)

50. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Apoptotic Index With PIC Once Daily for 21 Days (QD21D) Dosing
Description: as for outcome 46
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose and Days 7 and 21, 6 hours postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: apoptotic cells/millimeter of BEL
Arm/Group | Alisertib 25 mg PIC QD 21D | Alisertib 50 mg PIC QD 21D | Alisertib 70 mg PIC QD 21D
Number analyzed (Participants) | 3 | 6 | 7
apoptotic cells/millimeter of BEL
  Day 1, Hour 6: number analyzed (Participants) | 3 | 3 | 1
  Day 1, Hour 6 | 0.122 (0.2117) | 0.000 (0.0000) | 0.000 (NA) — Cannot be calculated for 1 participant
  Day 1, Hour 24: number analyzed (Participants) | 3 | 3 | 2
  Day 1, Hour 24 | 0.042 (0.0722) | 0.042 (0.0719) | 0.000 (0.0000)
  Day 7, Hour 6: number analyzed (Participants) | 0 | 0 | 3
  Day 7, Hour 6 |  |  | 0.000 (0.0000)
  Day 21, Hour 6: number analyzed (Participants) | 0 | 1 | 3
  Day 21, Hour 6 |  | 0.099 (NA) — Cannot be calculated for 1 participant. | 0.032 (0.0552)

51. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Mitotic Index With PIC Twice Daily for 7 Days (BID7D) Dosing
Description: as for outcome 45
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose and Day 7, 6 hours postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mitotic cells/millimeter of BEL
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 11 | 6
mitotic cells/millimeter of BEL
  Day 1, Hour 6: number analyzed (Participants) | 9 | 6
  Day 1, Hour 6 | 0.054 (0.3022) | 0.364 (0.2574)
  Day 1, Hour 24: number analyzed (Participants) | 6 | 6
  Day 1, Hour 24 | 2.578 (2.2875) | 1.435 (0.8329)
  Day 7, Hour 6: number analyzed (Participants) | 3 | 0
  Day 7, Hour 6 | 5.486 (5.8688) |

52. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Apoptotic Index With PIC Twice Daily for 7 Days (BID7D) Dosing
Description: as for outcome 46
Time Frame: Baseline and Cycle 1 Day 1, 6 hours and 24 hours postdose and Day 7, 6 hours postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: apoptotic cells/millimeter of BEL
Arm/Group | Alisertib 50 mg PIC BID 7D | Alisertib 60 mg PIC BID 7D
Number analyzed (Participants) | 11 | 6
apoptotic cells/millimeter of BEL
  Day 1, Hour 6: number analyzed (Participants) | 9 | 6
  Day 1, Hour 6 | -0.016 (0.0494) | 0.020 (0.0491)
  Day 1, Hour 24: number analyzed (Participants) | 6 | 6
  Day 1, Hour 24 | 0.055 (0.1691) | 0.080 (0.1958)
  Day 7, Hour 6: number analyzed (Participants) | 3 | 0
  Day 7, Hour 6 | 2.142 (3.2510) |

53. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Mitotic Index With PIC Twice Daily for 14 Days (BID14D) Dosing
Description: as for outcome 45
Time Frame: Baseline and Cycle 1 Day 7, 6 hours postdose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: mitotic cells/millimeter of BEL
Arm/Group | Alisertib 40 mg PIC BID 14D
Number analyzed (Participants) | 1
mitotic cells/millimeter of BEL | 1.507 (NA) — Cannot be calculated for 1 participant

54. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy as Measured by Apoptotic Index With PIC Twice Daily for 14 Days (BID14D) Dosing
Description: as for outcome 46
Time Frame: Baseline and Cycle 1 Day 7, 6 hours postdose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: apoptotic cells/millimeter of BEL
Arm/Group | Alisertib 40 mg PIC BID 14D
Number analyzed (Participants) | 1
apoptotic cells/millimeter of BEL | 2.837 (NA) — Cannot be calculated for 1 participant

55. Secondary Outcome: Number of Participants With Polymorphisms in Gene Encoding Enzyme UGT1A1
Description: One peripheral blood sample (approximately 4 mL) was to be obtained on Day 1 of Cycle 1 prior to the first dose of alisertib to genotype patients for polymorphisms in UGT1A1 because UGT1A1 is one of the enzymes responsible for glucuronidation of alisertib, which is expected to contribute to the clearance of alisertib.
  wt=wild type
  *28=polymorphism in the promoter region of a UGT1A1 allele resulting in reduced UGT1A1 expression.
Time Frame: Cycle 1 Day 1 predose
Population: Safety Population included all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Alisertib
Number analyzed (Participants) | 87
participants
  wt/wt | 38
  wt/*28 | 30
  *28/*28 | 9
  *28/other | 4
  other/other | 2
  Not Determined | 1
  Missing | 3

56. Secondary Outcome: Best Overall Response Based on Investigator Assessment
Description: Best overall response is defined as the percentage of participants with Complete Response (CR) + Partial Response (PR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1. According to RECIST: CR is defined as disappearance of all target and nontarget lesions and normalization of tumor marker level (if applicable); PR is defined as ≥30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter, persistence of 1 or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: Beginning at the end of Cycle 2, every 2 cycles until progressive disease (PD); Participants who discontinue study drug before PD: Follow-Up (FU) every 8-12 weeks until PD or as per institutional practice (Up to 33.2 months)
Population: Safety Population included all participants who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib
Number analyzed (Participants) | 87
percentage of participants | 1

57. Secondary Outcome: Duration Of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of a confirmed response to the date of first documented PD. PD is defined as 20% increase in the sum of the longest diameter of target lesions.
Time Frame: as for outcome 56
Population: Safety Population included all participants who received any amount of study drug.
Measure: Number; unit: days
Arm/Group | Alisertib
Number analyzed (Participants) | 1
days | 470

58. Secondary Outcome: Effect of Food on the Pharmacokinetics (PK) of Alisertib
Description: The effects of food on the PK of alisertib were to be evaluated using the preferred alisertib regimen (unit dose and formulation) based on the results from the relative bioavailability study.
Time Frame: Up to 6 months
Population: The effects of food on the PK of alisertib was not conducted. As the development of alisertib was transitioned from the PIC to the ECT formulation and the clinical dose of alisertib ECT had not been determined yet, it was decided that the effect of food would be evaluated in a different study at the appropriate clinical dose, administered as ECT.
Arm/Group | Alisertib 40 mg ECT BID 7D | Alisertib 40 mg PIC BID 7D
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last dose (up to 1011 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | PIC Dose Escalation | ECT Dose Escalation | Relative Bioavailability
Serious Adverse Events (participants affected / at risk) | 26/65 | 0/2 | 1/20
Other Adverse Events (participants affected / at risk) | 65/65 | 2/2 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PIC Dose Escalation (N=65) | ECT Dose Escalation (N=2) | Relative Bioavailability (N=20)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with alisertib 40 mg PIC BID14D (PIC dose escalation reporting group) and is not related.
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with alisertib 80 mg PIC QD7D (PIC dose escalation reporting group) and is not related.
Syncope (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with alisertib 40 mg PIC BID7D (PIC dose escalation reporting group) and is not related.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with alisertib 40 mg PIC QD7D (PIC dose escalation reporting group) and is not related.
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PIC Dose Escalation (N=65) | ECT Dose Escalation (N=2) | Relative Bioavailability (N=20)
Nausea (Gastrointestinal disorders) | 39 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 34 | 1 | 6
Vomiting (Gastrointestinal disorders) | 24 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 15 | 1 | 5
Constipation (Gastrointestinal disorders) | 12 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 13 | 0 | 2
Flatulence (Gastrointestinal disorders) | 5 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 0
Ascites (Gastrointestinal disorders) | 4 | 0 | 0
Oral pain (Gastrointestinal disorders) | 3 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 32 | 2 | 12
Oedema peripheral (General disorders) | 13 | 0 | 4
Pyrexia (General disorders) | 12 | 0 | 5
Asthenia (General disorders) | 11 | 1 | 1
Chills (General disorders) | 4 | 0 | 2
Gait disturbance (General disorders) | 3 | 0 | 1
Chest discomfort (General disorders) | 2 | 0 | 1
Pain (General disorders) | 1 | 1 | 1
Malaise (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 27 | 0 | 6
Dizziness (Nervous system disorders) | 13 | 0 | 3
Headache (Nervous system disorders) | 9 | 0 | 0
Paraesthesia (Nervous system disorders) | 6 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 28 | 0 | 7
Anaemia (Blood and lymphatic system disorders) | 24 | 2 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 30 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 9 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 1 | 10
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onychorrhexis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 21 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 6 | 0 | 1
Blood creatinine increased (Investigations) | 5 | 0 | 1
Weight decreased (Investigations) | 6 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 1
Platelet count decreased (Investigations) | 3 | 0 | 1
Weight increased (Investigations) | 3 | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 7 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 3
Confusional state (Psychiatric disorders) | 3 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2
Vision blurred (Eye disorders) | 4 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1
Visual disturbance (Eye disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Hepatobiliary disorders (Hepatobiliary disorders) | 4 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.